CLINICAL TRIAL: NCT06086327
Title: Chemokine Receptor CXCR4-targeting PET Imaging for Thymoma
Brief Title: Application of 68Ga-Pentixafor PET/CT for Thymoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-CXCR4-thymoma
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-06

CONDITIONS: Thymoma
MeSH Terms: conditions — Thymoma | interventions — 68Ga-pentixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-Pentixafor, PET/CT (Experimental): Inject 68Ga-Pentixafor and then perform PET/CT scan.
  Interventions: Drug: 68Ga-Pentixafor

INTERVENTIONS:
Drug: 68Ga-Pentixafor — Intravenous injection of one dosage of 74-185 MBq(2-5 mCi) 68Ga-Pentixafor. Tracer doses of 68Ga- Pentixafor will be used to image lesions of thymoma by PET/CT.
  Other Names: 68Ga-CXCR4

SUMMARY:
Chemokine receptor CXCR4 was expressed in T cells and CXCR4-targeting molecular imaging- 68Ga-Pentixafor PET/CT could be a promising technique to evaluate the extent of thymoma with higher accuracy. This prospective study is going to investigate whether metabolic characterization by 68Ga-Pentixafor PET/CT may be superior for diagnosis, distinguish evaluation for thymoma.

DETAILED DESCRIPTION:
Thymoma is 1 rare type of tumor developed on the thymic epithelium; patients with thymoma also might have myasthenia gravis (MG). Because of the scarcity and complexity of MG-associated thymoma, its pathogenesis and etiology still remain unclear nowadays. The expression of C-X-C chemokine receptor type 4 (CXCR4) is absent or low in most healthy tissues but highly expressed in various types of tumors. CXCR4 might contribute to the clinical cancer progression, and CXCR4 could be a valuable prognostic biomarker in the therapy of MG-associated thymoma.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed untreated thymoma patients
* signed written consent.

Exclusion Criteria:

* pregnancy
* breastfeeding
* known allergy against Pentixafor
* any medical condition that in the opinion of the investigator,may
* significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
SUVmax and SUVmean | through study completion, an average of 1.5 years
  SUVsof focal lesions are measured on 68Ga-Pentixafor PET/CT. The SUVs of the blood pool and muscle are defined as the background activity on the condition that there is no focally hypermetabolic disease.

SECONDARY OUTCOMES:
Diagnostic value | through study completion, an average of 1.5 years
  Diagnostic value of 68Ga-Pentixafor PET/CT for thymoma in comparison with 18F-FDG PET/CT or CT or MRI.
Diagnostic value in special type of thymoma | through study completion, an average of 1.5 years
  Diagnostic value of 68Ga-Pentixafor PET/CT in special type thymoma (A\AB\B\C subtypes)
Diagnostic value in thymoma and other masses | through study completion, an average of 1.5 years
  Diagnostic value of 68Ga-Pentixafor PET/CT in thymoma and other anterior mediastinal mass.
CXCR4 expression and SUV | through study completion, an average of 1.5 years
  Correlation between CXCR4 expression and SUV in PET

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospitall, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao X, Peng X, Wang R, Qian Z, Zhou X, Zhu Z, Chen Y. An Occult Primary Thymic Mucosa-Associated Lymphoid Tissue Lymphoma With Sjogren's Syndrome Revealed by CXCR4 Targeted 68Ga-Pentixafor PET/CT. J Cell Mol Med. 2025 Feb;29(3):e70248. doi: 10.1111/jcmm.70248. PMID 39887860